CLINICAL TRIAL: NCT00084448
Title: A Phase II Evaluation of Weekly Paclitaxel (NSC #673089) and Celecoxib (Celebrex®, NSC #719627) in the Treatment of Recurrent or Persistent Platinum-Resistant Epithelial Ovarian or Primary Peritoneal Cancer
Brief Title: Paclitaxel and Celecoxib in Treating Patients With Recurrent or Persistent Platinum-Resistant Ovarian Epithelial or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: GOG_0126P
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2005-06

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Celecoxib; Paclitaxel

INTERVENTIONS:
Drug: celecoxib
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may stop the growth of cancer by stopping blood flow to the tumor and may increase the effectiveness of paclitaxel by making tumor cells more sensitive to the drug. Giving celecoxib together with paclitaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel together with celecoxib works in treating patients with recurrent or persistent platinum-resistant ovarian epithelial or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of paclitaxel and celecoxib in patients with recurrent or persistent platinum-resistant ovarian epithelial or primary peritoneal cancer.
* Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and oral celecoxib twice daily on days 2-6, 9-13, and 16-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study within 11-22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or primary peritoneal cancer

  * Recurrent or persistent disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * At least 1 target lesion not in a previously irradiated field
* Must have received 1 prior platinum-based chemotherapy regimen for primary disease containing carboplatin, cisplatin, or another organoplatinum compound

  * Initial treatment may have included high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
  * Platinum-resistant or refractory (i.e., had a treatment-free interval after platinum therapy of less than 6 months OR disease progression during platinum-based therapy)
  * Patients who have not received a prior taxane may have received a second regimen that included paclitaxel or docetaxel
* Must not be eligible for a higher priority GOG protocol

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGOT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No neuropathy (sensory and motor) > grade 1
* No history of peptic ulcer disease
* No allergies to sulfa or non-steroidal anti-inflammatory drugs
* No known hypersensitivity to paclitaxel or celecoxib
* No other invasive malignancy within the past 5 years except non-melanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior biologic or immunologic therapy
* One prior non-cytotoxic* regimen for recurrent or persistent disease allowed NOTE: *Non-cytotoxic (biologic or cytostatic) agents include (but are not limited to) monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy
* No other prior cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial chemotherapy regimen

Endocrine therapy

* At least 1 week since prior hormonal therapy for malignant tumor
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* No prior radiotherapy to more than 25% of marrow-bearing areas

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* At least 3 weeks since prior therapy for malignant tumor
* No prior celecoxib
* No prior therapy for a previous cancer that would preclude protocol therapy
* No concurrent amifostine or other protective agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Antitumor activity
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte E. Miller, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa, United States